CLINICAL TRIAL: NCT02050867
Title: Validation of the Ask Suicide-Screening Questions (ASQ) in the Inpatient Medical Setting
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: Boston Children's Hospital (Other); Children's National Research Institute (Other); Nationwide Children s Hospital in Columbus, Ohio (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914044; 14-M-N044
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09-12

CONDITIONS: Children; Adolescents
Keywords: Youth Suicide; Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Physicians and nurses working in non-mental health settings require tools to guide them in recognizing patients at risk. While screening children and adolescents is emerging as a priority of the Joint Commission, there are currently no suicide screening instruments designed specifically for assessing suicide risk in a pediatric inpatient medical population. Recently, our study team developed the Ask Suicide-Screening Questions (ASQ), a 4-item suicide risk screening instrument with excellent sensitivity, specificity, and negative predictive value for use in pediatric emergency departments (Protocol #08-M-N070). However, use of the ASQ in an inpatient medical setting has not been tested. The aim of this study is to determine the utility of the ASQ among pediatric medical inpatients in children s hospitals. While most inpatients will not be at imminent risk for suicide, we hypothesize that the ASQ will capture a number of patients who screen positive and are not only at risk for suicidal behavior in the future, but are also experiencing significant emotional distress and therefore warrant further psychiatric evaluation and follow-up treatment. This will be a multisite study, comprised of medically ill inpatients at three non-NIH affiliated sites (Children s National Medical Center, Boston Children s Hospital, and Nationwide Children s Hospital), with a total sample size of 600 (200 per site). We will administer several short measures of suicide risk the ASQ, the Suicidal Ideation Questionnaire, a brief depression screen, the Patients Health Questionnaire Adolescent version (PHQ-A) to all eligible inpatients aged 10-21 years. The ultimate goal of this project is to provide non-mental health clinicians with a brief, accurate assessment tool for detecting risk of suicide in pediatric medical inpatients and in turn, connecting those in need with mental health services. After validating the ASQ with pediatric medical inpatients, we will then examine the practical implications of nurses administering the ASQ as standard of care during the admission process on a pediatric medical inpatient unit. Future studies will focus on validating the ASQ in non-English speaking patients, addressing a critical gap in suicide prevention research. In addition, examining the long-term clinical impact of screening general medical patients for suicide risk with the ASQ and linking those in need with mental health services and/or other interventions will be important next steps.

Please note: This is a multi-site study that is being conducted at three non-NIH sites, all children s hospitals, two of which have already received IRB approval (Boston Children s Hospital and Children s National Medical Center) and one which is in the process of submission (Nationwide Children s Hospital). No NIH patients will be enrolled at the Clinical Center. Consent and patient data collection will take place on inpatient medical units at those three sites; data will be sent to NIMH, and stored and analyzed here.

DETAILED DESCRIPTION:
Physicians and nurses working in non-mental health settings require tools to guide them in recognizing patients at risk. While screening children and adolescents is emerging as a priority of the Joint Commission, there are currently no suicide screening instruments designed specifically for assessing suicide risk in a pediatric inpatient medical population. Recently, our study team developed the Ask Suicide-Screening Questions (ASQ), a 4-item suicide risk screening instrument with excellent sensitivity, specificity, and negative predictive value for use in pediatric emergency departments (Protocol #08-M-N070). However, use of the ASQ in an inpatient medical setting has not been tested. The aim of this study is to determine the utility of the ASQ among pediatric medical inpatients in children s hospitals. While most inpatients will not be at imminent risk for suicide, we hypothesize that the ASQ will capture a number of patients who screen positive and are not only at risk for suicidal behavior in the future, but are also experiencing significant emotional distress and therefore warrant further psychiatric evaluation and follow-up treatment. This will be a multisite study, comprised of medically ill inpatients at three non-NIH affiliated sites (Children s National Medical Center, Boston Children s Hospital, and Nationwide Children s Hospital), with a total sample size of 600 (200 per site). We will administer several short measures of suicide risk the ASQ, the Suicidal Ideation Questionnaire, a brief depression screen, the Patients Health Questionnaire Adolescent version (PHQ-A) to all eligible inpatients aged 10-21 years. The ultimate goal of this project is to provide non-mental health clinicians with a brief, accurate assessment tool for detecting risk of suicide in pediatric medical inpatients and in turn, connecting those in need with mental health services. After validating the ASQ with pediatric medical inpatients, we will then examine the practical implications of nurses administering the ASQ as standard of care during the admission process on a pediatric medical inpatient unit. Future studies will focus on validating the ASQ in non-English speaking patients, addressing a critical gap in suicide prevention research. In addition, examining the long-term clinical impact of screening general medical patients for suicide risk with the ASQ and linking those in need with mental health services and/or other interventions will be important next steps.

Please note: This is a multi-site study that is being conducted at three non-NIH sites, all children s hospitals, all of which have already received IRB approval (Boston Children s Hospital, Children s National Medical Center and Nationwide Children s Hospital). The CNS IRB requires that we have an NIMH parent protocol even though no NIH patients will be enrolled at the Clinical Center. Consent and patient data collection will take place on inpatient medical units at those three sites; data will be sent to NIMH, and stored and analyzed here.

ELIGIBILITY:
* INCLUSION CRITERIA:<TAB>

All pediatric medical inpatients, aged 10 to 21 years, who are current inpatients on selected medical units at the three different sites during data collection weeks, will be approached for enrollment. Patients will be included if: 1) they are admitted as an inpatient from Sunday at 7am through Thursday 11:59pm and 2) they have a parent or legal guardian who is present to sign informed consent (for patients under 18 years of age)

EXCLUSION CRITERIA:<TAB>

Patients will be excluded if: 1) they have severe developmental delays, cognitive impairment, or communication disorder such that the patient is not able to comprehend questions or communicate their answers; 2) their illnesses are so severe that the study staff feels that they may not able to comprehend questions or communicate their answers; 3) they have primarily psychiatric disorders and are boarding ; 4) parents/guardians

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 562 (Actual)
Dates: Start 2014-01-29; Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures include frequencies of positive responses to all ASQ and SIQ items. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Horowitz, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Childrens Hospital, Columbus, Columbus, Ohio, United States

REFERENCES:
- [Background] Furlanetto LM, Stefanello B. Suicidal ideation in medical inpatients: psychosocial and clinical correlates. Gen Hosp Psychiatry. 2011 Nov-Dec;33(6):572-8. doi: 10.1016/j.genhosppsych.2011.08.002. Epub 2011 Sep 9. PMID 21908051
- [Background] Qin P, Webb R, Kapur N, Sorensen HT. Hospitalization for physical illness and risk of subsequent suicide: a population study. J Intern Med. 2013 Jan;273(1):48-58. doi: 10.1111/j.1365-2796.2012.02572.x. Epub 2012 Aug 12. PMID 22775487
- [Background] Christiansen E, Stenager E. Risk for attempted suicide in children and youths after contact with somatic hospitals: a Danish register based nested case-control study. J Epidemiol Community Health. 2012 Mar;66(3):247-53. doi: 10.1136/jech.2009.103887. Epub 2010 Oct 14. PMID 20947873
- [Derived] Horowitz LM, Wharff EA, Mournet AM, Ross AM, McBee-Strayer S, He JP, Lanzillo EC, White E, Bergdoll E, Powell DS, Solages M, Merikangas KR, Pao M, Bridge JA. Validation and Feasibility of the ASQ Among Pediatric Medical and Surgical Inpatients. Hosp Pediatr. 2020 Sep;10(9):750-757. doi: 10.1542/hpeds.2020-0087. PMID 32826283
- [Derived] Ross AM, White E, Powell D, Nelson S, Horowitz L, Wharff E. To Ask or Not to Ask? Opinions of Pediatric Medical Inpatients about Suicide Risk Screening in the Hospital. J Pediatr. 2016 Mar;170:295-300. doi: 10.1016/j.jpeds.2015.11.052. Epub 2015 Dec 24. PMID 26725208